CLINICAL TRIAL: NCT04196855
Title: Study of Teriparatide in Stress Fracture Healing
Acronym: RETURN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of East Anglia (Other)
Collaborators: Ministry of Defence, United Kingdom (Other Government); Darlington Memorial Hospital (Unknown); Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19/HRA/6011
Record Dates: First submitted 2019-12-05; First posted 2019-12-12 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2019-12

CONDITIONS: Stress Fracture; Parathyroid Hormone
MeSH Terms: conditions — Fractures, Stress | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded assessment of MR scans
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention - Teriparatide Treatment (Experimental): Teriparatide 20ug/day from confirmation of stress fracture for 16 weeks, with the potential to extend to 24 weeks if required.
  Interventions: Drug: Teriparatide
- Control - Standard Care (No Intervention): Standard rehabilitation care with additional monitoring to assess healing.

INTERVENTIONS:
Drug: Teriparatide — Terrosa 20 micrograms/80 microliters solution for injection. Each dose of 80 microliters contains 20 micrograms of teriparatide.
  One cartridge of 2.4 mL of solution contains 600 micrograms of teriparatide (corresponding to 250 micrograms per mL).
  Teriparatide, rhPTH(1-34), produced in E. coli, using recombinant DNA technology, is identical to the 34-N-terminal amino acid sequence of endogenous human parathyroid hormone.
  Other Names: Terossa
  Arms: Intervention - Teriparatide Treatment

SUMMARY:
Investigation into the use of teriparatide in the treatment of stress fractures.

Primary outcome is healing on MRI, secondary outcomes are pain, time spent in rehabilitation and future stress fractures. This study will help the investigators understand how to treat stress fractures in the future.

DETAILED DESCRIPTION:
Teriparatide is a drug that is designed to have a similar effect on the body as parathyroid hormone. Parathyroid hormone is made naturally in the body and is released in response to low calcium levels. It helps to maintain bone health and repair bone damage. Parathyroid hormone and medicines like teriparatide can strengthen bones and are often given to people with osteoporosis (a condition that weakens bones, making them more likely to break) to reduce the risk of fractures. Recent studies have also shown benefits in people with stress fracture injuries, a form of bone damage sometimes caused by repetitive exercise. The investigators want to know if teriparatide is also beneficial to healthy, younger people who have a stress fracture injury.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form;
2. Participant must be aged 18 - 40 years inclusive;
3. Participant must have a lower limb stress fracture, either unilateral or bilateral, as confirmed via MRI scan;
4. Undergoing phase 1 or 2 training within an Army training establishment;
5. Blood Tests within reference range. Minor abnormalities will be assessed by the PI. Patients will still be entered if these are felt to be of no clinical importance.
6. Participants able to adhere to the visit schedule and protocol requirements.

Exclusion Criteria:

1. Hypersensitivity to the active Parathyroid Hormone substance or any of the excipients listed in the SmPC.
2. Pre-existing hypercalcaemia.
3. Patients with skeletal malignancies or bone metastases.
4. Any contraindications that would prevent the participant from undergoing an MRI scan.
5. Concurrent therapy that, in the investigators opinion, would interfere with the evaluation of the safety or efficacy of the study medication.
6. Pregnancy, suspected pregnancy or breastfeeding. Female participants must have a negative serum pregnancy test at screening and be willing and able to use a "highly effective" method of contraception, as per the Clinical Trial Facilitation Group (CTFG) guidance.
7. Severe renal impairment. Participants with moderate renal impairment will be treated with caution at the Principal Investigator's discretion and in accordance with the SmPC.
8. Metabolic bone diseases including hyperparathyroidism and Paget's disease of the bone.
9. Unexplained elevations of alkaline phosphatase.
10. Prior external beam or implant radiation therapy to the skeleton.
11. Patients participating in a concurrent drug trial.
12. Presentation with open epiphyses during the diagnostic MRI scan.
13. Participants with depression, as identified by completion of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Baseline.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2019-12-23 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Radiological healing. | 8 weeks.
  Radiological healing by 2 Grades or more, or to grade zero at 8 weeks.

SECONDARY OUTCOMES:
Radiological Healing | 8, 10, 12, 14, 16, 20, 24 weeks
  Time to complete radiological healing
Time from randomisation to assessed as 'Clinically Healed'. | Twice weekly from date of radiologically healed stress fracture reported on MRI scan up to 24 weeks
  Physical assessment to commence once the fracture is reported as healed on MR.
Time to 'Healing' as a composite assessment. | Up to 24 weeks.
  Healing as assessed by MRI and clinical assessment.
Time from randomisation to discharge from rehabilitation. | Up to 24 weeks
  Completion of rehab will be assessed using Army standard measures.
Pain symptoms on a visual analogue pain scale. | Diary to be completed weekly and analysed as a change from baseline to 16 weeks (24 weeks in an unhealed fracture).
  Score between 0 and 10 - with 0 being no pain and 10 being worst pain imaginable.
Difference in Quality of life | 4 weekly from baseline to 16 weeks
  Assessed by Short Form 36 Questionnaire. The higher score, the better the participants quality of life.
Adverse events | Up to 28 weeks.
  As reported in accordance with CTAE Version 4.03

OTHER OUTCOMES:
P1NP response to teriparatide treatment. | Base line then 4 weekly to week 16 - extorted to week 24 in the case of an unhealed fracture.
  Measurement of bone marker of formation.
CTX response to teriparatide treatment. | Base line then 4 weekly to week 16 - extorted to week 24 in the case of an unhealed fracture.
  Measurement of bone marker of formation.

CONTACTS AND LOCATIONS:
Overall Officials: William Fraser, Dr, Principal Investigator — Norwich Medical School
Locations (1):
- Darlington Memorial Hospital, Darlington, County Durham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carswell AT, Eastman KG, Casey A, Hammond M, Shepstone L, Payerne E, Toms AP, MacKay JW, Swart AM, Greeves JP, Fraser WD. Teriparatide and stress fracture healing in young adults (RETURN - Research on Efficacy of Teriparatide Use in the Return of recruits to Normal duty): study protocol for a randomised controlled trial. Trials. 2021 Aug 30;22(1):580. doi: 10.1186/s13063-021-05556-3. PMID 34461961